CLINICAL TRIAL: NCT07232043
Title: AI-driven Clinical-trial Trial-Information and Viability Assessment Tool for EHRs (ACTIVATE)
Brief Title: ACTIVATE: AI-driven Clinical-trial Trial-Information and Viability Assessment Tool for EHRs
Acronym: ACTIVATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kenneth Kehl, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-413; 1R37CA295653-01A1 (NIH)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Cancer; Clinical Trial Enrollment; Electronic Health Records; Artificial Intelligence
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard MatchMiner-AI Workflow (No Intervention): Oncologists can access the MatchMiner-AI frontend website to obtain a list of clinical trial options for all participants.
- Proactive AI-Triggered Notifications (Experimental): Oncologists receive email notifications containing a ranked list of potential clinical trial options when AI models detect progressive disease, in addition to standard MatchMiner-AI access.
  Interventions: Other: MatchMiner-AI Artificial Intelligence Tool

INTERVENTIONS:
Other: MatchMiner-AI Artificial Intelligence Tool — Oncologists receive email notifications containing a ranked list of potential clinical trial options when AI models detect progressive disease, in addition to standard MatchMiner-AI access.
  Other Names: MatchMiner-AI Pipeline
  Arms: Proactive AI-Triggered Notifications

SUMMARY:
This study aims to develop and evaluate ACTIVATE, an AI-driven tool for clinical trial information and viability assessment using electronic health records (EHRs). The project will leverage retrospective and prospective EHR data to build and validate algorithms that identify potentially eligible participants for clinical trials and facilitate trial matching.

DETAILED DESCRIPTION:
ACTIVATE is a pragmatic health system intervention designed to improve clinical trial matching and accrual using AI-driven tools integrated with EHR data. The study will first retrospectively analyze data from approximately 70,000 participants who initiated new systemic therapy at Dana-Farber Cancer Institute since 2016 to develop and validate the MatchMiner-AI pipeline.

For the prospective evaluation, all DFCI patients' medical record numbers (MRNs) will be randomized into control and intervention groups. The intervention group will receive proactive notifications to treating oncologists when AI models detect progressive disease and a high probability of starting new treatment, including a ranked list of potential clinical trial options. The control group will continue with standard MatchMiner-AI workflows.

ELIGIBILITY:
Inclusion Criteria:

* 3.1 The potentially eligible patient population includes any adult (≥18 years old) with a cancer diagnosis receiving care at DFCI. No direct patient recruitment will occur as part of this protocol; all data will be obtained retrospectively or prospectively from routine clinical documentation and electronic health records. TrialForecast will involve aggregate queries of this dataset for cohort size estimation. The randomized interventional component (TrialMatch) is a health system level email "nudge" to treating oncologists providing a list of clinical trial options for patients who have progressive disease based on their imaging reports as detected using our previously developed, validated, and deployed AI model for that purpose. 23-25 Secondary outcomes in our study will include oncologist satisfaction with information delivered via these pipelines. All DFCI oncologists at any DFCI-owned/operated site (Longwood, Chestnut Hill, and regional campus sites) will be eligible to use our pipeline and may receive notifications about clinical trial options for their patients. In 2024, there were approximately 593 such oncologists who had outpatient appointments with at least one patient. Clinicians will constitute study participants as well, since they will have the opportunity to provide feedback on our pipeline to be analyzed by the study team.
* 3.2 Our project will focus on adults with cancer treated at DFCI, as above. We will not have any mechanism for identifying, targeting, or excluding pregnant women or prisoners.

Exclusion Criteria:

* 3.2 Our project will focus on adults with cancer treated at DFCI, as above. We will not have any mechanism for identifying, targeting, or excluding pregnant women or prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion clinical trials | Assessment will occur at the end of the 1.5 year duration of the intervention.
  The effect of TrialMatch notifications is defined as the proportion of new systemic therapy starts which are clinical trials.

SECONDARY OUTCOMES:
Proportion clinical trials by race | Assessment will occur at the end of the 1.5 year duration of the intervention.
  The effect of TrialMatch notifications is defined as the proportion of new systemic therapy starts which are clinical trials. The outcome will be stratified by race categories of: American Indian/Alaska Native, Asian, Native Hawaiian or Other Pacific Islander, Black or African America, White, and More than One Race.
Proportion clinical trials by ethnicity | Assessment will occur at the end of the 1.5 year duration of the intervention.
  The effect of TrialMatch notifications is defined as the proportion of new systemic therapy starts which are clinical trials. The outcome will be stratified by ethnicity (Hispanic or non-Hispanic)
Proportion clinical trials by age | Assessment will occur at the end of the 1.5 year duration of the intervention.
  The effect of TrialMatch notifications is defined as the proportion of new systemic therapy starts which are clinical trials. The outcome will be stratified by Age categories of: 18-29 years, 30-39 years, 40-49 years, 50-59 years, 60-69 years, 70-79 years, 80-89 years, and 90+ years.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Kehl, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: kenneth_kehl@dfci.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu